CLINICAL TRIAL: NCT06374316
Title: Air Purifiers in Classrooms for Infection Control - a Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: SINTEF Health Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2302888
Record Dates: First submitted 2024-01-30; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-02

CONDITIONS: Feasibility; Acceptability
Keywords: Infection Control; Air Purifier; Covid-19; School
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: We will select schools for participation in arm 1 and 2, respectively, based on the feasibility of installing ceiling-mounted and placing portable air purifiers in each relevant classroom. In arm 3, all three classrooms will be equipped with both ceiling-mounted and portable air purifiers, as well as indoor air quality sensors.
  For this arm, we will randomize the three classrooms to each of three weekly programs for the air purifiers;
  Program 1) Week 1, 4, and 7: Ceiling-mounted ON, Week 2, 5, and 8: No purifier on, Week 3, 6, and 9: Portable ON. Program 2) Week 1, 4, and 7: Portable ON, Week 2, 5, and 8: Ceiling-mounted ON, Week 3, 6, and 9: No purifier on. Program 3) Week 1, 4, and 7: No purifier on Week 2, 5, and 8: Portable ON, Week 3, 6, and 9: Ceiling-mounted ON.
  Each classroom will be assigned a computer-generated random number and will based on the ascending order of the random numbers be allocated to the three predetermined sequences of programs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ceiling-Mounted Air Purifiers (Experimental): Classrooms in this arm will have ceiling-mounted air purifiers installed. Air quality will be monitored throughout the study period.
  Interventions: Device: Ceiling-Mounted Air Purifiers
- Portable Air Purifiers (Experimental): Classrooms in this arm will have portable air purifiers installed. Air quality will be monitored throughout the study period.
  Interventions: Device: Portable Air Purifiers
- Both Portable and Ceiling-Mounted Air Purifiers (Experimental): Classrooms in this arms will have both portable and ceiling-mounted air purifiers installed. The rooms will alternate weekly between having no air purifiers on, or only ceiling-mounted air purifier on, or only portable air purifier on.
  Air quality will be monitored throughout the study period.
  Interventions: Device: Portable or Ceiling Mounted Air Purifiers

INTERVENTIONS:
Device: Ceiling-Mounted Air Purifiers — The devices will be turned on every working day except Tuesdays. Air purifiers will be set at levels perceived as acceptable by both teachers and students during operational hours.
  Arms: Ceiling-Mounted Air Purifiers
Device: Portable Air Purifiers — The devices will be turned on every working day except Tuesdays. Air purifiers will be set at levels perceived as acceptable by both teachers and students during operational hours.
  Arms: Portable Air Purifiers
Device: Portable or Ceiling Mounted Air Purifiers — The Ceiling-Mounted and Portable devices will alternate weekly between being activated and deactivated in the three classrooms. Each classroom will also have three weeks with no purifier activated.This alternating pattern aims to assess the impact of the various air purifiers on air quality. Air purifiers will be set at levels perceived as acceptable by both teachers and students during operational hours.
  Arms: Both Portable and Ceiling-Mounted Air Purifiers

SUMMARY:
This study aims to investigate the acceptability and feasibility of deploying air purifiers equipped with HEPA (high-efficiency particulate air) filters in classrooms, to study air purifiers as an infection control measure. It will also evaluate the direct effect of air purifiers on air quality, comparing ceiling-mounted purifiers, portable purifiers and no purifier.

DETAILED DESCRIPTION:
Improved ventilation and air purification have been proposed as promising measures to protect the health of students and children while avoiding future school closures during pandemics. However, there is limited knowledge regarding the effectiveness and potential drawbacks of using air purifiers in educational settings. This pilot study was initiated to explore whether a large study of air purifiers in Norwegian primary school classrooms is feasible and acceptable among teachers and students, and to uncover whether air purifiers can reduce particle density in classrooms and thus potentially decrease the spread of infections.

The results will lay the groundwork for larger-scale trials that could form the basis of knowledge for decision-makers on whether the use of air purifiers should be part of the strategy to limit infections in classrooms while avoiding school closures during future pandemics.

The pilot study consists of two parts. The first part will last six weeks, and focus on the feasibility and acceptability among teachers and students. It will describe and compare two arms - ceiling-mounted (arm 1) and portable (arm 2) air purifiers. The second part lasts nine weeks, and will evaluate the direct effect of air purifiers on air quality. It will compare ceiling-mounted, and portable devices and no purifier(arm 3). The study will involve multiple schools, with a total of six schools contributing eight classrooms. Arm 1 will have two schools and arm 2 will have three schools, each school contributing with one classroom. Arm 3 will have one school, contributing with three classrooms. The classrooms will preferably belong to 7th grade students, but 6th and 5th grade student classrooms will also be accepted, based on the schools preferences. Data collection includes interviews and questionnaires from teachers and students, observations, as well as absenteeism data and air quality measurements.

ELIGIBILITY:
Inclusion Criteria for Schools in arm 1 and 2:

* Having a classroom in the 5th to 7th grade that either has sufficient floor space to accommodate at least two portable air purifiers or has the infrastructure for the installation of a ceiling-mounted air purifier.
* Having at least 15 students in the relevant classroom.

Inclusion Criteria for Schools in arm 3:

* Having three classrooms at the same floor with sufficient floor space to accommodate at least two portable air purifiers AND with the infrastructure for the installation of a ceiling-mounted air purifier.
* The relevant three classrooms should be slightly comparable with regards to use and air quality. The air quality, as perceived by users, should generally be rated as moderate to poor. which should be medium to poor.

Inclusion Criteria for Students in arm 1 and 2:

* Having a classroom with installed air purifier through the study as their primary classroom.
* Informed consent from both legal guardians.

Inclusion Criteria for Teachers in arm 1, 2, and 3:

* Teaching in the classroom with installed air purifiers at least a few hours per week.
* Providing informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of air purifiers versus no air purifier on improving air quality in classrooms. | 9 weeks
  Air quality will be measured using specialized monitors, capturing key indicators such as particulate matter levels. The data collected will enable a comprehensive evaluation of the effectiveness of air purifiers versus no air purifier in improving the overall air quality in educational settings.
Effectiveness of ceiling mounted versus portable air purifier on improving air quality in classrooms. | 9 weeks
  Air quality will be measured using specialized monitors, capturing key indicators such as particulate matter levels. The data collected will enable a comprehensive evaluation of the effectiveness between ceiling mounted and portable air purifiers in improving the overall air quality in educational settings.
Acceptability of having Air Purifiers in Classrooms | 6 weeks
  Acceptability will be assessed through the in-depth qualitative interviews with teachers and students, exploring perceptions and challenges associated with the use of air purifiers.
Untoward events when installing air purifiers in classrooms | 2 weeks
  Experiences will be collected from the personnel involved in installing the air purifiers
Untoward events when running air purifiers in classrooms | 9 weeks
  Experiences will be collected from class teachers and students through in-depth qualitative interviews at the beginning (only teachers) and the end (teachers and students) of the study period. Observations and experiences from the study team during the study period will be collected and described.
How student absence data can be collected from existing school registration systems. | 8 weeks
  Experiences from collecting data from the individual schools or from the municipalities, on absence per week per class based on the existing absence systems, will be described.

SECONDARY OUTCOMES:
Response rate of class teachers to the study surveys. | 6 weeks
  Consent will be sought from relevant teachers in part 1 schools, and weekly questionnaires will be sent out. Response rates will be described. Results will be supported by answers to interview questions about motivations and challenges in participating in such surveys.
Response rate of students/their guardians to study surveys. | 8 weeks
  Consent will be sought from students in part 1 schools, and weekly questionnaires will be sent out. Response rate will be described.
Proportion of absence due to respiratory disease. | 8 weeks
  Answers to surveys from teachers and students on absence and reasons for absence, from part 1 schools, will be analysed.
Absence frequency among students | 8 weeks
  Based on the absence data from the schools existing registration systems, we will describe the absence frequency among students in the participating classes.

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

REFERENCES:
- See also: Study Protocol — https://zenodo.org/records/10526802